CLINICAL TRIAL: NCT06428656
Title: The Effect of Postbiotics Supplementation on Gut Microbiota Composition and Exercise-induced Inflammation
Brief Title: Postbiotics Supplementation, Gut Microbiota Composition, and Exercise-induced Inflammation
Acronym: PostBioExIn
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Chariklia K. Deli, Associate Professor, University of Thessaly
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Screening
Other Study IDs: PB-GM-Exercise-Inflammation
Record Dates: First submitted 2024-05-20; First posted 2024-05-24 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Postbiotics Supplementation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The randomization of the participants to the supplement or placebo condition will be performed via a random integer set generator (Random.org) available online.
  Neither the participants, nor the care provider, nor the investigator will be aware of whether participants receive the postbiotic supplement or the placebo. Additionally, blood samples will be masked during the biochemical analysis, and during the statistical analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Postbiotics supplementation (Experimental): Supplementation of postbiotics for 4 weeks
  Interventions: Dietary Supplement: Postbiotics supplementation
- Placebo supplementation (Placebo Comparator): Supplementation of placebo for 4 weeks
  Interventions: Dietary Supplement: Placebo supplementation

INTERVENTIONS:
Dietary Supplement: Postbiotics supplementation — The participants will consume one capsule of postbiotics supplement per day
  Arms: Postbiotics supplementation
Dietary Supplement: Placebo supplementation — The participants will consume one capsule of placebo per day
  Arms: Placebo supplementation

SUMMARY:
This study will investigate the effect of postbiotics supplementation on gut microbiota (GM) composition, exercise-induced oxidative stress and performance following eccentrically biased exercise. The study will be a cross-over, randomized, double-blind, controlled study that will be conducted in two cycles. Participants will be randomly assigned into one of the two trials: i) Postbiotics supplementation for 4 weeks, ii) Placebo supplementation for 4 weeks. Participants will then perform a 45-min treadmill running at (-15% slope, ~70% VO2max) followed by a time-trial (0% slope, ~95% VO2max) until exhaustion. Before, as well as 24 h, 48 h and 72 h following exercise, assessment of GM composition and metabolites (short-chain fatty acids), exercise induced muscle damage (EIMD) (delayed onset of muscle soreness, creatine kinase), complete blood count (CBC), blood inflammatory status (tumor necrosis factor alpha, interleukin 6, C-reactive protein), gut inflammatory status (lipopolysacharides-binding protein, zonulin), blood redox status (total antioxidant capacity, catalase, protein carbonyls, reduced glutathione, oxidized glutathione, and performance (knee-extensors' and knee-flexors' isometric, concentric, eccentric torque, countermovement jump) will be performed. In addition, metabolism (lactic acid) will be assessed before and 4 min following exercise. Afterwards, the participants will receive the postbiotics supplement or the placebo for 4 weeks, and will repeat the exercise protocol and measurements of EIMD, CBC, blood inflammatory status, blood redox status and performance at the same time-points. At the second cycle, the participants will repeat the above procedures under the remaining condition. Between conditions, there will be a 14-day washout period. The results of the research will provide important information for coaches and physically active individuals, regarding the effectiveness of postbiotics to favorably change the gut microbiota composition and alleviate gut inflammation, exercise-induced inflammation and oxidative stress, and improve performance after intense exercise.

DETAILED DESCRIPTION:
Acute, vigorous and/or unaccustomed eccentric exercise can induce muscle injury and inflammatory reactions, and oxidative stress, but also reduced muscle performance. For this reason, many professional as well as amateur athletes, often consume nutritional supplements such as antioxidants, anticipating to reduce inflammation and oxidative stress after intense exercise.

The human gastrointestinal tract is inhabited by various microorganisms, called the gut microbiome (GM). GM, among other things, contributes to the normal functioning of the immune system, contributes to the production of short-chain fatty acids (SCFAs) and vitamin synthesis as well as the digestion and absorption of food, protects against enteropathogens and regulates inflammatory and redox responses. Recent evidence also suggests that GM may be involved in athletic performance. In contrast, disruption of GM composition (dysbiosis) is characterized by reduced diversity, reduced abundance of health-promoting bacteria, and increased abundance of gram-negative and other pathogenic bacteria and is associated with various metabolic diseases such as obesity, diabetes, and various forms of cancer, systemic inflammation, oxidative stress and reduced performance. Thus, the supplementation of several "biotics" has been emerged as a means to regulate the GM in favor of health-promoting bacteria.

Postbiotics is defined as a "preparation of inanimate microorganisms and/or their components that confers a health benefit on the host". Evidence suggests that supplementation with postbiotics may regulate the GM, and consequently, strengthen the immune system, reduce intestinal permeability, improve antioxidant mechanisms, as well as accelerate recovery after exercise-induced inflammation, enhance adaptations to exercise, and improve performance. However, the scientific data regarding the possible beneficial effect of supplemental administration of postbiotics is limited. More research is needed, in order to determine the role of postbiotics supplementation on GM composition and function, exercise-induced inflammation and redox status, but also on performance after intense exercise.

This study will investigate the potential of postbiotics supplementation to alter the GM composition and affect the recovery of exercise-induced oxidative stress and performance following intense, eccentrically biased acute exercise. The study will be cross-over, randomized, double-blind, controlled, and will be conducted in two cycles. The participants, will be primarily informed regarding the study procedures, as well as the benefits and possible risks, and will sign an informed consent form for participation in the study. Before the experimental procedure, they will be involved in a week of familiarization to the evaluation tests and the exercise protocol, at a low intensity. Participants will undergo baseline measurements: anthropometric characteristics (body height, body mass, body mass index) via a stadiometer-scale (Stadiometer 208; Seca, Birmingham, UK), body composition (amount of body fat, lean body mass, fat mass, bone density) via by dual emission X-ray absorptiometry (DXA, GE-Healthcare, Lunar DPX NT, Belgium), aerobic capacity (VO2max) via an automated online pulmonary gas analyzer (Vmax Encore 29, BEBJO296, Yorba Linda, CA, USA) during a graded exercise protocol on a treadmill (Stex 8025T, Korea), isokinetic strength (isometric, concentric and eccentric torque of the knee extensors and knee flexors) on an isokinetic dynamometer (Cybex, HUMAC NORM 360, Ronkonkoma, NY), and muscle power via the assessment of countermovement jump (CMJ) via an optical measurement system (Optojump next, Microgate, USA). In addition, the participants will record their diet via a 7-days recall before their participation in the first experimental condition, and dietary data will be analyzed with ScienceFit Diet 200A diet analysis program (Science Technologies, Athens, Greece), in order to estimate that they do not consume nutrients that may affect muscle injury, inflammation and oxidative stress (e.g. antioxidants, etc.). Participants will then be randomized in one of the two conditions: i) Postbiotics supplementation (50mg/day of Heatkilled Lactobacillus plantarum L-137, Immuno-LP20TM) for 4 weeks, or ii) placebo supplementation for 4 weeks. Randomization of the conditions will be done by a software generating random integers available on the internet (Random.org). Participants will then perform an exercise protocol comprised of 45 min downhill running (-15% slope, ~70-75% VO2max) on a treadmill followed by a time-trial (0% slope, ~95% VO2max) until exhaustion. Before the exercise protocol, as well as 24 h, 48 h and 72 h after exercise, exercise-induced muscle damage (EIMD) [delayed onset of muscle soreness (DOMS) via palpation of the knee extensors and knee flexors on a scale of 1 to 10 (1 = no pain at all; 10 = extreme pain), and muscle performance (CMJ, isometric, concentric and eccentric torque of the knee extensors and knee flexors)], will be assessed. At the same time points, feces samples will be collected for the analysis of GM composition and function, and GM metabolites, as well as blood samples for the assessment of complete blood count (CBC), blood inflammatory status (creatine kinase, tumor necrosis factor alpha, interleukin 6, C-reactive protein), gut inflammatory status (lipopolysacharides-binding protein, zonulin), and blood redox status [reduced glutathione (GSH), oxidized glutathione (GSSG), GSH/GSSG ratio, total antioxidant capacity, catalase, protein carbonyls, uric acid, bilirubin). Furthermore, metabolism (lactic acid) will be assessed before and 4 min following exercise by analyzing capillary blood with a portable lactate analyzer (Lactate Plus, Nova Biomedical, USA). Afterwards, the participants will receive the postbiotics supplement or the placebo for 4 weeks, and will repeat the exercise protocol and measurements of EIMD, CBC, blood inflammatory status, blood redox status and performance at the same time-points. At the second cycle, participants will repeat the exact same procedures for the remaining condition. Between cycles, a 14-days washout period will be applied. Additionally, the 7-day diet recall from the first cycle, will be given to the participants to follow the same diet before the experimental exercise protocol at the second cycle.

ELIGIBILITY:
Inclusion Criteria:

* Physically active subjects (VO2max ≥35ml/kg/min)
* Absence of musculoskeletal injury (≥6 months)
* Abstinence from the use of ergogenic supplements (≥1 month)
* Abstinence from anti-inflammatory drugs (≥1 month)
* Abstinence from pre-pro-postbiotic supplements (≥6 months)
* Abstinence from participating in exercise with eccentric content for at least 7 days before exercise
* Abstinence from alcohol and energy drinks before exercise

Exclusion Criteria:

* Recent history of musculoskeletal injury (<6 months)
* Use of ergogenic performance supplements (<1 month)
* Taking anti-inflammatory drugs (<1 month)
* Taking pre-pro-postbiotic supplements (<6 months)
* Participation in exercise with eccentric content in the previous 7 days before exercise
* Consumption of alcohol and energy drinks before exercise

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Changes in gut microbiota composition | At baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-exercise
  Gut microbiota composition will be assessed in feces
Changes in butyrate | At baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-exercise
  Butyrate will be assessed in feces
Changes in propionate | At baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-exercise
  Propionate will be assessed in feces
Changes in acetate | At baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-exercise
  Acetate will be assessed in feces
Changes in complete blood count | At baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-exercise
  Complete blood count will be assessed in whole blood
Changes in creatine kinase activity | At baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-exercise
  Creatine kinase activity will be assessed in serum
Changes in TNF-α concentration | At baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-exercise
  TNF-α concentration will be assessed in serum
Changes in IL-6 concentration | At baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-exercise
  IL-6 concentration will be assessed in serum
Changes in high-sensitivity C-reactive protein concentration | At baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-exercise
  C-reactive protein concentration will be assessed in serum
Changes in lipopolysacharides-binding protein concentration | At baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-exercise
  Lipopolysacharides-binding protein concentration will be assessed in serum
Changes in zonulin concentration | At baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-exercise
  Zonulin concentration will be assessed in serum and in feces
Changes in protein carbonyls concentration | At baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-exercise
  Protein carbonyls concentration will be assessed in plasma
Changes in malondialdehyde concentration | At baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-exercise
  Malondialdehyde concentration will be assessed in plasma
Changes in reduced glutathione concentration | At baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-exercise
  Glutathione concentration will be assessed in red blood cells lycate
Changes in oxidized glutathione concentration | At baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-exercise
  Oxidized glutathione concentration will be assessed in red blood cells lycate
Changes in GSH/GSSG ratio | At baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-exercise
  GSH/GSSG ratio will be assessed in red blood cells lycate
Changes in catalase concentration | At baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-exercise
  Catalase concentration will be assessed in red blood cells lycate
Changes in total antioxidant capacity | At baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-exercise
  Total antioxidant capacity will be assessed in red blood cells lycate
Changes in uric acid concentration | At baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-exercise
  Uric acid concentration will be assessed in serum
Changes in bilirubin concentration | At baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-exercise
  Bilirubin concentration will be assessed in serum
Changes in blood lactate concentration | At baseline (pre), 4 min post-exercise
  Bilirubin concentration will be assessed in whole blood
Changes in delayed onset of muscle soreness in the knee flexors and extensors of both limbs | At baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-exercise
  Muscle soreness of the KF and KE will be assessed via palpation of the muscle belly and the distal regions following 3 squats, and the subjective pain will be recorded on a 10-point scale (1 = no pain, 10 = extreme pain)
Changes in countermovement jump height | At baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-exercise
  Countermovement jump height will be measured with an optical system
Changes in isokinetic strength of knee extensors and knee flexors | At baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-exercise
  Isometric, concentric and eccentric peak torque of the knee extensors and knee flexors of both limbs will be assessed on an isokinetic dynamometer

CONTACTS AND LOCATIONS:
Overall Officials: Chariklia K Deli, PhD, Principal Investigator — University of Thessaly
Locations (1):
- Department of Physical Education and Sport Science, Uninersity of Thessaly, Trikala, Thessaly, Greece